CLINICAL TRIAL: NCT03096106
Title: The Reliability and Validity of Visual Assessment for Pressure-time Curve
Brief Title: Visual Assessment for Pressure-time Curve
Status: Completed | Type: Observational
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jian-Xin Zhou, Professor, Capital Medical University
Other Study IDs: KY2017-016-02
Record Dates: First submitted 2017-03-16; First posted 2017-03-30 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-03

CONDITIONS: Mechanical Ventilation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device:  — the investigators just observe the pressure time curve on the ventilation

SUMMARY:
Airway pressure-time (P-t) curve and stress index (SI) assessment have been proposed to guide the mechanical ventilation settings and minimize ventilator-induced lung injury.

DETAILED DESCRIPTION:
The stress index (SI), which has been proposed to guide the mechanical ventilation settings and minimize ventilator-induced lung injury. It reflects the change of respiratory compliance during inspiration. Value of SI equals to 1 that indicates a constant compliance, whereas values lower and higher than 1 indicate increase and decrease of compliance over inspiratory time, suggesting tidal recruitment and tidal hyperinflation, respectively. Based on the different values of SI showing different shapes, SI of straight curve equals to 1, SI of concave curve lower than 1 and convex curve higher than 1, the investigators speculated that the SI value could be reliably and accurately estimated by visual inspection of the P-t curve.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older; intubated and mechanical ventilated by volume-control ventilation with constant flow;

Exclusion Criteria:

* evidence of active air leak from the lung, including bronchopleural fistula, pneumothorax, pneumomediastinum, or existing chest tube; evidence of the stiff chest wall, such as existing the pleural effusion, intra abdominal hypertension, chest injuries and abdominal injuries.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: intubated and mechanical ventilated by volume-control ventilation with constant flow
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
the types of pressure time curve by visual inspection. | up to 10min, from the ventilator screen being frozen to the two observers completing judgement.
  the pressure time curves have the three types:the straight,concave,convex,the observers will judge the types of pressure time curve by visual inspection, and record the results of judgement

CONTACTS AND LOCATIONS:
Overall Officials: Jian-xin zhou, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- ICU, Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun XM, Chen GQ, Chen K, Wang YM, He X, Huang HW, Luo XY, Wang CM, Shi ZH, Xu M, Chen L, Fan E, Zhou JX. Stress Index Can Be Accurately and Reliably Assessed by Visually Inspecting Ventilator Waveforms. Respir Care. 2018 Sep;63(9):1094-1101. doi: 10.4187/respcare.06151. Epub 2018 Jun 26. PMID 29945907